CLINICAL TRIAL: NCT05028803
Title: The Effects of Sodium Phenylbutyrate on Circulating Branched Chain Amino Acid Concentrations in Obese and Prediabetics.
Brief Title: The Effects of Sodium Phenylbutyrate on Circulating Branched Chain Amino Acids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Philip Atherton, Professor Philip athertone, University of Nottingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: _COMAP; 135-1220 (Other: University of Nottingham)
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Obese Non Diabetic
MeSH Terms: interventions — 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phenylbutyrate (Experimental): Volunteers will recieve 5 grams of Sodium Phenylbutyrate daily for 3 weeks (21 days). Sodium Pheburane will come in granuale form and 5 grams will be dosed every day.
  Interventions: Drug: sodium phenylbutyrate

INTERVENTIONS:
Drug: sodium phenylbutyrate — same as arm/group

SUMMARY:
The aim of this study is to reduce fasting circulating BCAA concentrations in volunteers using Sodium Phenylbutyrate. In addition, we aim investigate the effect of BCAA lowering on fasting blood glucose levels, insulin sensitivity measures and muscle metabolism.

DETAILED DESCRIPTION:
A total of twenty proteinogenic amino acids are present in the human body1. Due to their chemical structure, three of the amino acids - isoleucine, leucine and valine, are termed branched chain amino acids (BCAAs). Humans consume BCAAs through protein containing foods such as meat, eggs and milk2,3. However, recent studies, have revealed links between elevated plasma levels of BCAAs and type 2 diabetes (T2D), insulin resistance (IR) and obesity4-6. Such is the strength of these links that elevated blood concentration of BCAAs are considered biomarkers and prognostic factors for obesity, insulin resistance and type 2 diabetes7-9. Collectively, these data suggest that targeting dysregulation of BCAAs by reducing BCAA levels could offer important therapeutic value. Various methods can be implemented in order to reduce circulating fasting BCAA concentrations one method that our department has successfully implemented includes the restriction of BCAAs in 6 healthy volunteer participants through diet control. By restricting BCAA in the diets of healthy individuals, we successfully reduced fasting circulating BCAAs by 50% in just seven days. However, the construction of the diet was very time consuming, tedious, and longer studies would be plagued with compliance issues. This has led us to try an alternative method, which is to lower BCAA levels using Sodium Phenylbutyrate (NaPB). NaPB is a commonly used medication to treat patients with urea cycle disorders (UCD). However, it seems a secondary effect of the drug is to reduce circulating BCAA levels in volunteers. Lindsey Burrage et al 2014, reported significantly lower circulating BCAAs in volunteers receiving NaPB when compared to subjects not receiving NaPB10. Although the mechanisms are not fully understood it has been suggested that NaPB causes depletion of glutamine in the blood which may activate BCAA catabolism and thus cause a reduction in circulating plasma BCAAs11. It is our aim to use NaPB to lower BCAAs in prediabetic and obese participants.

Screening Visit Volunteers will sign a consent form, A health assessment, including an ECG to monitor your heart, a blood pressure check, height and weight measurement and a medical history check A fasted blood sample to measure health parameters, including glucose, HbA1c, liver and kidney function, lipid profiles, thyroid function and full blood count.

Once we received the details and results (within 1 week) from your screening session, we will contact you regarding your suitability. If you are suitable, we (you and the research team together) will decide on the dates to start the programme.

Instruct you in the completion of a food diary. STUDY DAY 0 For this day, we will ask volunteers to attend after an overnight fast (except water). We will take small samples of your blood (fasting sample).

After the blood samples participants will receive a 'heavy water' drink called Deuterium Oxide (D2O). This is almost the same as normal water, but a small and harmless chemical change allows us to calculate how much new muscle your body is making. The amount of D2O you are given will be calculated based on your body weight. Participants will provide saliva samples before and after receiving D2O. Before they go home they will receive small daily top-ups of D2O and asked to collect your saliva 3 hours after taking your daily top-ups for the first week, and twice weekly thereafter and keep the saliva samples in a fridge/freezer.

STUDY DAY 7 On return for the second study day participants will also bring with them saliva samples from the last 7 days. For this day, again volunteers are to attend after an overnight fast (except water). We will perform a muscle biopsy (fasting sample) to use as our baseline/pre-intervention measures. A fully qualified medical practitioner will take muscle biopsies. Biopsies are sterile procedures, with local anaesthetic.

Muscle biopsies Muscle biopsies will be taken from the thigh. Before the biopsy, the area will be cleaned and anaesthetised with local anaesthetic, after which a small (approx. 1cm wide, 2-3cm deep) incision will be made through the skin. The muscle biopsy (smaller than the size of a pea) will then be removed from the thigh using conchotome forceps (essentially a sharp pair of tweezers), with 3-5 small pieces taken to ensure adequate sampling. The incision will then be stitched shut and covered with a waterproof adhesive dressing. Muscle biopsies are usually well tolerated, largely painless (though the insertion is felt) and the complication rate is very low.

Biopsy Aftercare At the end of the biopsy, you will receive advice and information about how to take care of the wound and given an information leaflet. Five to seven days after each muscle biopsy, the stitches will be removed and the wounds will be checked.

In addition to the above, volunteers will also have a series of minimally and non-invasive tests to assess different aspects of your health and metabolic status:

1. We will measure how well the body is able to process sugar by performing the oral glucose tolerance test (OGTT). This is usually used to diagnose diabetes, or stratify the future risk of diabetes. For this test, you will be given 75g of a sugary drink. Small blood samples will be taken prior to the drink and every 15 minutes (for 2 hours) from a cannula (thin plastic line) sited in a vein in your hand, which will be placed in a warm box.
2. A light lunch will be provided at midday. After lunch the first oral dose of phenyl butyrate will be given.
3. Volunteers will receive the first dose of Phenylbutyrate after lunch. Volunteers will receive 5 grams of sodium Phenylbutyrate every day. 5 g/m2/day of Sodium Phenylbutyrate will be split into three and taken with each meal.
4. Participants will receive Sodium Phenylbutyrate to last one week. STUDY DAY 10 For this day, we will ask you to attend after an overnight fast (except water). We will take small samples of your blood (fasting sample). In addition, blood pressure, weight and height will be recorded. Volunteers will also have an ECG. It is anticipated study day 11 will take up to 1 hour to complete.

STUDY DAY 17 For this day, we will ask you to attend after an overnight fast (except water). We will take small samples of your blood (fasting sample) and a saliva sample to use as our midpoint intervention measures. In addition, blood pressure, weight and height will be recorded. Volunteers will then be provided with another medication organiser box with enough Sodium Phenylbutyrate to last them until the end of the study. It is anticipated study day 17 will take up to 1 hour to complete. We will also request a test for Leukopenia.

STUDY DAY 28 This is the final day of the study, again volunteers are to attend after an overnight fast (except water). A fully qualified medical practitioner will take muscle biopsies. Biopsies are sterile procedures, with local anaesthetic. Following this, we will perform the oral glucose tolerance test (OGTT), volunteers will be given 75g of a sugary drink. Small blood samples will be taken prior to the drink and every 15 minutes (for 2 hours) from a cannula which will be placed in a warm box In addition, blood pressure, weight and height will also be recorded. In addition a Fructosamine test will also be requested pre and post study.

ELIGIBILITY:
Inclusion Criteria:

* • Participant is willing and able to give informed consent for participation in the study

  * Not currently taking any medications
  * Males between the ages of 18 - 60
  * BMI ≥ 30 kg·m2
  * FBG ≥ 6 mmol/L ≤ 7mmol/L or HbA1c ≥ 42 mmol/mol 48 ≤ mmol/mol

Exclusion Criteria:

* • Specify any diseases/disorders/ conditions that would preclude entry into the study

  * Females
  * History or current psychiatric illness
  * History or current neurological condition (e.g. epilepsy)
  * Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance (this must remain for ALL UoN FMHS UREC approved studies)
  * A BMI < 30kg·m2
  * FBG >7mmol/L/ or HbA1c >48mmol/mol
  * Metabolic disease; Active inflammatory bowel disease
  * Chronic kidney disease
  * Malignancy
  * Recent (6 mo) steroid/ hormone therapy
  * Clotting dysfunction
  * Musculoskeletal/ neurological disorders
  * Active cardiovascular disease or recent cardiac event
  * Respiratory disease (not including well-controlled asthma)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Serum branched chain amino acids (BCAA) levels | 3 weeks
  Both total and individual BCAAs before and after intervention

SECONDARY OUTCOMES:
Musle protein syntyhesis (MPS) | 4 weeks
  Estimation via weekly sampling of saliva following deuterium oxide (D2O) tracer solution administration relative to baseline.
Metabolic status (Oral glucose tolerance testing (OGTT)) | 3 weeks
  Undertaken to assess for insulin sensitivity and resistance.

OTHER OUTCOMES:
Glycated haemoglobin (Hba1c) glucose metabalism testing via venepuncture | 3 weeks
  Assessment of Hba1c pre and post intervention-results are compared against local laboratory reference range.
Fructosamine glucose metabalism testing via venepuncture | 3 weeks
  Assessment of fructosamine pre and post intervention-results are compared against local laboratory reference range.
Immune statis (full blood count via venepuncture) | 3 weeks
  Frequent monitoring of full blood count lebvels to asess for leukopenia. Results are compared against local laboratory refernec range, pre, peri and post study.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Prof Athertone, DM, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant medical information obtained as a result of this study are considered confidential and disclosure to third parties is prohibited with the exceptions noted above. Such medical information may be given to the participant's medical team and all appropriate medical personnel responsible for the participant's welfare. If information is disclosed during the study that could pose a risk of harm to the participant or others, the researcher will discuss this with the Chief Investigator (CI) and where appropriate report accordingly. Data generated as a result of this trial will be available for inspection on request by the participating physicians, the University of Nottingham representatives, the local Research Ethics Committee (REC) and the regulatory authorities. Elements of the results from this study will be submitted for peer-review in at least one publication.